CLINICAL TRIAL: NCT07154095
Title: A Single-Center, Randomized, Open-Label, Two-Sequence, Two-Period, Crossover Study to Compare the Pharmacokinetics and Safety of Pyridostigmine Sustained-Release Tablets and Pyridostigmine Tablets Following Single and Multiple Doses in Healthy Chinese Participants
Brief Title: A Single-Center, Randomized, Open-Label, Two-Sequence, Two-Period, Crossover Study Comparing the Pharmacokinetics and Safety of Pyridostigmine Sustained-Release and Immediate-Release Tablets Following Single and Multiple Doses in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Yu Qin, West China Second University Hospital, West China Second University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CRC-C2142
Record Dates: First submitted 2025-08-25; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Myasthenia Gravis; Pharmacokinetics
MeSH Terms: conditions — Myasthenia Gravis | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Intervention Model Description: A single-center, randomized, open-label, two-sequence, two-period, crossover design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sustained-release pyridostigmine tablet (Experimental)
  Interventions: Drug: Sustained-Release Tablets
- Immediate-Release Tablets (Active Comparator)
  Interventions: Drug: Immediate-Release Tablets

INTERVENTIONS:
Drug: Sustained-Release Tablets — A single-center, randomized, open-label, two-sequence, two-period, crossover design was employed. Forty healthy participants were enrolled and randomized (1:1) into two sequences (AB and BA) to receive both the test and reference formulations across two periods, separated by a washout interval of at least 5 days.
  Arms: sustained-release pyridostigmine tablet
Drug: Immediate-Release Tablets — A single-center, randomized, open-label, two-sequence, two-period, crossover design was employed. Forty healthy participants were enrolled and randomized (1:1) into two sequences (AB and BA) to receive both the test and reference formulations across two periods, separated by a washout interval of at least 5 days.
  Other Names: MESTINON®
  Arms: Immediate-Release Tablets

SUMMARY:
This study aimed to assess the pharmacokinetic profile, safety, and tolerability of a new sustained-release pyridostigmine tablet versus the reference product. The evaluation was conducted in healthy participants following both single and multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 45 years (inclusive), male or female;
2. Weight: male ≥50 kg, female ≥45 kg; body mass index (BMI) within the range of 19-26 kg/m² (inclusive);
3. Normal or abnormal without clinical significance in physical examination, vital signs, 12-lead electrocardiogram (ECG), laboratory tests, and chest X-ray;
4. Negative test results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), and Treponema pallidum antibody;
5. No plans for childbearing or sperm/egg donation during the trial and for 3 months after the last dose, and willingness to use reliable contraceptive measures;
6. Ability to communicate well with the researchers, fully understand the purpose of the trial, comply with all requirements, voluntarily participate in the clinical trial, and provide written informed consent.

Exclusion Criteria:

1. Known history of allergy to the investigational drug or any of its components, or related preparations; history of allergic diseases or allergic constitution;
2. History of any disease that may affect the safety of the participant or the pharmacokinetics of the investigational drug, including but not limited to central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematopoietic system, metabolic disorders (e.g., hyperkalemia), or other conditions unsuitable for clinical trials (e.g., psychiatric history), or history of mechanical intestinal obstruction, urinary tract obstruction, or bronchial asthma;
3. Chronic excessive consumption (more than 8 cups per day, 1 cup = 250 mL) of tea, coffee, or caffeine-containing beverages; or intake of any food or beverage containing caffeine, grapefruit, or poppy seeds (e.g., coffee, alcohol, strong tea, chocolate, grapefruit, pomelo, etc.) within 48 hours prior to the first dose;
4. Difficulty in blood collection or inability to comply with a standardized diet;
5. History of blood donation (including component blood donation) or blood loss ≥ 200 mL, or receipt of blood transfusion within 3 months prior to the first dose;
6. Smoking ≥10 cigarettes per day;
7. Positive alcohol breath test, or regular alcohol consumption (exceeding 21 units per week, 1 unit containing 14 g of alcohol, e.g., 360 mL of beer, 45 mL of 40% spirits, or 150 mL of wine) within 3 months prior to the first dose;
8. History of drug abuse or drug dependence, or positive urine drug abuse screening (morphine, tetrahydrocannabinol, methamphetamine, methylenedioxymethamphetamine, ketamine);
9. Use of any prescription drugs, herbal tonics, or any drugs that inhibit or induce liver drug metabolism within 1 month prior to the first dose, and/or use of any over-the-counter drugs or dietary supplements (including vitamins, calcium tablets, etc.) within 2 weeks prior to the first dose;
10. Participation in any other clinical trial and receipt of an investigational drug within 3 months prior to the first dose;
11. Lactating females or those with a positive pregnancy test (applicable to female participants);
12. Other factors deemed by the investigators to be unsuitable for participation in the trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Tmax | Blood sampling: Within 1 hour pre-dose and 24 hours post-dose on Day 1; within 5 to 2 minutes pre-dose and 24 hours post-dose on Day 5.
  Time to Reach Maximum Concentration
Cmax | Blood sampling: Within 1 hour pre-dose and 24 hours post-dose on Day 1; within 5 to 2 minutes pre-dose and 24 hours post-dose on Day 5.
  Peak Concentration
AUC | Blood sampling: Within 1 hour pre-dose and 24 hours post-dose on Day 1; within 5 to 2 minutes pre-dose and 24 hours post-dose on Day 5.
  Area under the plasma concentration-time curve

SECONDARY OUTCOMES:
TEAE | From first dose of study drug up to a maximum of 6 days
  Treatment-emergent adverse event (TEAE): any adverse event that first appears or worsens in severity after initiation of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yu Qin, Principal Investigator — China West China Second University Hospital Chengdu, China
Locations (1):
- West China Second University Hospital, Chengdu, China